CLINICAL TRIAL: NCT00619463
Title: Effects of Aerobic Exercise on Cognition, Mood and Fatigue Following TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1R49CE001171-01 (NIH)
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Exercise; Cognition; Brain Derived Neurotrophic Factor (BDNF); peripheral vascular endothelial growth factor (VEGF)
MeSH Terms: conditions — Brain Injuries, Traumatic; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise then monitor (Experimental): 8 weeks of aerobic exercise followed by 16 weeks of monitoring
  Interventions: Behavioral: Exercise
- monitor than exercise (Experimental): 8 weeks of monitoring followed by 16 weeks of aerobic exercise
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Eight weeks in an aerobic exercise program- 50 minutes of aerobic exercise on a treadmill - 3 days a week for 8 -16 weeks.
  Arms: exercise then monitor
Behavioral: Exercise — Aerobic exercise program - 55 min aerobic exercise on the treadmill 3 days a week for either 8 or 16 weeks
  Arms: monitor than exercise

SUMMARY:
The purpose of the study is to determine the efficacy of aerobic exercise for improving cognition, mood, and fatigue after Traumatic Brain Injury (TBI) as well as examine the role of Brain Derived Neurotropic Factor (BDNF) and peripheral Vascular Endothelial Growth Factor (VEGF) as mediators of response to exercise.

DETAILED DESCRIPTION:
The cognitive, emotional and physical effects of TBI are well documented in the literature. Specifically, reduced cognitive functioning and depression, which are much more prevalent than in the general population, represent key challenges in the rehabilitation of persons recovering from TBI. Aerobic exercise has been shown to improve cognition and mood in the general population. Although the positive effects of exercise have been known for some time, only recently have some of the mechanisms underlying these effects been defined. One hypothesized mechanism was that exercise elevates the levels of BDNF and VEGF in the CNS. Although research examining the effects of aerobic exercise in individuals with TBI is limited, exercise has been effective in improving cognition and depression in individuals with other medical conditions, such as cancer, multiple sclerosis, fibromyalgia, dementia, chronic fatigue syndrome, chronic obstructive pulmonary disease and the elderly.

The effects of aerobic exercise on patients with TBI will be examined in this clinical trial, using a crossover design with a wait-list control. The classic crossover design has been modified to examine the effects of an additional 8 weeks of exercise, for a total 16-week intervention, in one group. Participants will be randomized into one of two conditions: Group A - immediate eight weeks of intervention followed by monitoring or Group B - monitoring followed by 8 weeks of intervention. In addition, the participants in Group B will serve as their own controls to determine if another 8 weeks of exercise, for a total of 16 weeks, is necessary for cognitive improvement.

Each person will undergo individual interviews and testing/ questionnaires aimed at measuring cognition, mood, fatigue, and life satisfaction. Blood will be drawn 2 or 3 times to monitor BDNF and VEGF levels. Assessment of cognition, mood, fatigue and life satisfaction will occur at four time points for both groups.

It is hypothesized that aerobic exercise will result in improved cognition and mood from both subjective and objective perspectives. In addition, we will explore the effect of post-TBI exercise on community participation and life satisfaction and explore personal and injury characteristics that mediate effectiveness of aerobic exercise in individuals with TBI.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 to 99
* Have experienced a TBI as a result of a blow to the head with a loss of consciousness or a period of being dazed and confused. This must be medically documented (e.g. EMS report, hospital record, physician record).
* Be at least six-months post-injury
* Be English-speaking since assessments and treatment sessions will be conducted by English-speaking therapists
* Have residential telephone service since follow up assessments may be completed via phone
* Live within 1.5 hours of NYC to be able to participate in baseline assessment and attend treatment sessions
* Provide written informed consent for participation
* Be willing to complete questionnaires and interviews about mood, thinking skills, fatigue, and life satisfaction
* Being willing to comply with protocol requirements and a schedule of exercise and assessments visits
* Being able to take part in a treadmill-based exercise program

Exclusion Criteria:

* Any medical condition in which exercising may be harmful, e.g., evidence of cardiovascular compromise including: history of acute myocardial infarction, history of coronary artery disease, unstable angina, uncontrolled hypertension, orthostatic hypotension, significant aortic valve disease, uncontrolled arrhythmia, uncompensated congestive heart failure, 3rd degree AV block without a pacemaker, active pericarditis, active myocarditis, or any evidence of pulmonary, endocrine or neurologic compromise; impaired left ventricular dysfunction; or syncopal episode within the past year
* Any medical condition requiring treatment with beta blockers or calcium channel blockers
* Under the age of 18 years of age
* Any clinically significant evidence of pulmonary, endocrine or neurologic (ataxia, gait disturbance, vertigo) compromise
* Resting pulse oxymetry of less than 95% oxygen (O2) saturation, in normal air
* Recent diagnosis of deep vein thrombosis or pulmonary embolism
* Active systemic illness or chronic infection that is not stable
* Active inflammatory process that is not stable
* Clinically significant anemia
* Clinically significant abnormal thyroid function tests
* Pregnant females
* Any reason that, in the investigator's opinion, makes the person unsuitable to participate
* Unable to physically participate in an exercise program
* Active participation in regular aerobic exercise in the six months prior to potential enrollment.
* Active substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2007-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Hopkins Verbal Learning Test-Revised (HVLT-R) | Every 8 weeks for 24 weeks
Trail Making Tests A and B (TMT) | Every 8 weeks for 24 weeks
Digit span subtests of the WAIS-III | Every 8 weeks for 24 weeks
Wisconsin card sort test (WCST) | Every 8 weeks for 24 weeks
Controlled Oral Word Association Test (COWAT) | Every 8 weeks for 24 weeks
Stroop Word Color Test | Every 8 weeks for 24 weeks
Global Fatigue Index (GFI) | Every 8 weeks for 24 Weeks.
Beck Depression Inventory-II ( BDI-II) | Every 8 weeks for 24 Weeks.
Blood draws for assessment of BDNF and VEGF levels | Every 8 weeks for 24 weeks

SECONDARY OUTCOMES:
Injury characteristics and demographic variables | At the beginning of the study. Week 1 of 24
BISQ - Brain Injury Screening Questionnaire | At the beginning of the study. Week 1 of 24
Life 3 | Every 8 weeks for 24 Weeks
Transition Measures | Every 8 weeks for 24 Weeks
University of Rhode Island Change Assessment (URICA) | Every 8 weeks for 24 Weeks
Exercise Diaries | Once a day
International Physical Activity Questionnaire (IPAQ) | Once a week

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Gordon, Ph.D., Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States